CLINICAL TRIAL: NCT00457990
Title: Early Versus Late Enteral Iron Supplementation in Infants With a Birth Weight of Less Than 1301g - Neurocognitive Development at 5.3 Years Corrected Age
Brief Title: Neurodevelopment After Early Iron Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: UL-NEO-IRON-2
Record Dates: First submitted 2007-04-06; First posted 2007-04-09 (Estimated); Last update posted 2007-04-09 (Estimated); Status verified 2007-04

CONDITIONS: Iron Deficiency; Anemia of Prematurity; Neurodevelopmental Delay
Keywords: Neurocognitive outcome; preterm infant; very low birth weight; iron deficiency; iron supplementation
MeSH Terms: conditions — Iron Deficiencies; Anemia; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Oral administration of ferrous sulphate

SUMMARY:
Background: Iron deficiency in early childhood may impair neurodevelopment.

Aim: To examine whether early iron supplementation improved neurodevelopment in preterm infants.

Method: Children who participated in a clinical trial of iron supplementation were invited for a neurodevelopmental follow-up examination at the time of school entry.

DETAILED DESCRIPTION:
Children with a birth weight of < 1301g who participated in a randomized controlled trial of early versus late enteral iron supplementation were evaluated applying a standardized neurological evaluation, the Kaufmann Assessment Battery for Children, and the Gross Motor Function Classification Scale (GMFCS) at the age of school entry.

Severe disability was defined as any of the following: any abnormal neurological examination associated with a severely impaired mobility (GMFCS>1), severe cognitive impairment (mental processing composite (MPC) <51), hearing loss requiring amplification, or blindness. The absence of disability was defined as normal neurological examination, normal mobility (GMFCS=0), and normal cognitive development (MPC>85) and the absence of any severe hearing and visual impairment.

ELIGIBILITY:
Inclusion Criteria:

* inborn infants with a birth weight of <1301g admitted between June 1996 and June 1999

Exclusion Criteria:

* major anomalies, hemolytic disease, twin-to-twin transfusion syndrome, missing parental consent

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 204
Dates: Start 2002-04; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
ferritin at 61 days of life
the number of infants who fulfilled the criteria of ID at any time throughout the study.

SECONDARY OUTCOMES:
Neurological Status
Mental Processing Composite (Kaufmann Assessment Battery for Children)
Disability Status
Behavioural Problems

CONTACTS AND LOCATIONS:
Overall Officials: Axel R Franz, MD, Principal Investigator — University of Ulm
Locations (1):
- University Children's Hospital, Ulm, Germany

REFERENCES:
- [Derived] Steinmacher J, Pohlandt F, Bode H, Sander S, Kron M, Franz AR. Randomized trial of early versus late enteral iron supplementation in infants with a birth weight of less than 1301 grams: neurocognitive development at 5.3 years' corrected age. Pediatrics. 2007 Sep;120(3):538-46. doi: 10.1542/peds.2007-0495. PMID 17766527